CLINICAL TRIAL: NCT03488927
Title: Development and Pilot Trial of an Intervention to Reduce Disclosure Recipients Negative Social Reactions and Victims Psychological Distress and Problem Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Hampshire (Other)
Collaborators: University of Illinois at Chicago (Other); University of South Florida (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Katie Edwards, Associate Professor of Psychology, University of New Hampshire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNewHampshire
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Social Skills; Self-Criticism; Post-traumatic Stress Disorder; Depression; Alcohol Abuse; Drinking, College; Alcohol Drinking; Alcohol; Harmful Use; Social Stigma; Social Norms; Social Responsibility; Social Behavior; Empathy; Coping Skills; Coping Behavior
Keywords: Sexual Violence; Interpersonal Violence; Prevention; Mixed-Methods; Randomized Controlled Trial; Outcome Evaluation; College Students; Post-traumatic Stress Disorder; Alcohol; Sexual Assault; Disclosure; Social Reactions; Coping; Depression; Intervention
MeSH Terms: conditions — Social Skills; Stress Disorders, Post-Traumatic; Depression; Alcoholism; Alcohol Drinking in College; Alcohol Drinking; Social Stigma; Social Behavior

STUDY DESIGN:
Intervention Model Description: Randomized control intervention trial with a wait-list control condition, randomized at the individual level
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will receive the intervention, followed by a six-month follow-up evaluation.
  Interventions: Behavioral: Supporting Survivors and Self: An Intervention for Social Supports of Survivors of Partner Abuse and Sexual Aggression (SSS)
- Wait-list Control (No Intervention): This arm will receive the intervention after a six-month follow-up evaluation.

INTERVENTIONS:
Behavioral: Supporting Survivors and Self: An Intervention for Social Supports of Survivors of Partner Abuse and Sexual Aggression (SSS) — The SSS intervention consists of a two-hour session followed by a 90-minute booster session a month following the initial program session. The SSS intervention is delivered in groups of approximately 20 students facilitated by peer educators. The SSS intervention provides participants with specific information on the reasons why positive social reactions are important and negative social reactions can be harmful, examples of what to say and what not to say (including ways to promote healthy coping and discourage unhealthy coping, e.g., drinking to cope), opportunities for roleplay, and an emphasis on the importance of self-care and ways in which self-care can be balanced with the needs of IPV and SA victims.
  Arms: Intervention

SUMMARY:
The purpose of this randomized controlled trial is to evaluate an intervention, Supporting Survivors and Self: An Intervention for Social Supports of Survivors of Partner Abuse and Sexual Aggression (SSS). SSS trains potential recipients of IPV or SA disclosure on the best methods of responding to a victim's disclosure. Consenting college students will be randomized into the SSS intervention or a wait-list control condition. Evaluation data will be multi-informant (i.e., data from both informal supports and victims) and multi-method (i.e., qualitative and quantitative). The investigators hypothesize that individuals receiving the SSS intervention, compared to individuals in the wait-list control condition, will provide less negative and more positive social reactions to victims' disclosure.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) and sexual assault (SA) are public health issues that impact the vast majority of college students in some capacity (as a victim and/or disclosure recipient). Most (75+%) victims disclose to informal supports, such as friends. Unfortunately, over 80% of victims' disclosures are met with negative social reactions (e.g., blame) from informal supports (used interchangeably with disclosure recipients). Negative social reactions predict deleterious psychological (e.g., posttraumatic stress disorder) and behavioral (e.g., problem drinking) health outcomes in victims. Although recent research has shed light on the factors (e.g., victim attributions) that predict informal supports' negative (e.g., egocentric and blaming statements) and positive (e.g., providing emotional support) social reactions, there is no intervention to date that targets potential recipients of IPV and SA disclosure to inform these individuals of the best methods of responding to an IPV or SA disclosure. This type of intervention, if effective in reducing negative social reactions in informal supports, could reduce problem drinking and related outcomes in victims.

Thus, in the current study, the investigators evaluate an intervention (i.e., Supporting Survivors and Self [SSS]) created for potential informal support disclosure recipients. College students are the target population for the initial version of the SSS intervention given the high rates of SA, IPV, and alcohol misuse among this demographic. The interactive, two-session intervention teaches potential disclosure recipients what to say and not to say and ways to promote healthy coping and discourage unhealthy coping in victims. The role of alcohol in risk for and outcomes associated with IPV and SA as well as alcohol-specific social reactions are addressed in the SSS intervention because alcohol is involved in most situations of IPV and SA among college students, and drinking to cope is common among victims.

This study is a small-scale, yet rigorous, initial evaluation of the SSS intervention that includes a prospective (i.e., intervention prior to potential disclosure) and experimental (i.e., randomized control trial) methodology. Outcome data will be multi-informant (i.e., data from both informal supports and victims) and multi-method (i.e., qualitative and quantitative). The investigators will:

1. Implement and evaluate the effectiveness of the SSS intervention compared to a wait-list control condition among potential informal supports. Hypothesis 1a: Individuals receiving the SSS intervention (N=450) compared to individuals in the wait-list control condition (N=450) will report fewer IPV and SA rape myths as well as greater intentions to provide positive social reactions and fewer intentions to provide negative social reactions. Hypothesis 1b: Individuals who receive SSS intervention and are subsequent disclosure recipients (n=100) will report providing less negative social reactions and more positive social reactions than individuals in the control condition who are subsequent disclosure recipients (n=100); mediators (e.g., low victim blame) and moderators (e.g., victim alcohol use at time of assault) of outcomes will be examined. Hypothesis 1c: Individuals who receive the SSS intervention and are subsequent victims of IPV and/or SA (n=60) will report less self-blame, PTSD, depression, drinking to cope, and problem drinking compared to individuals in the control condition who are subsequent victims of IPV and/or SA (n=60); mediators (e.g., engagement in healthy coping) and moderators (e.g., gender) will be explored. Methodology: A random sample of college students from a public university will be invited to participate in a pre-test (all participants), SSS intervention (only participants randomly assigned to this condition), and six-month post-test (all participants). A subsample of disclosure recipients in the SSS intervention condition will be invited to participate in a qualitative exit interviews (after the post-test) to enrich findings and inform SSS revisions.
2. Determine the feasibility in recruiting victims who disclosed to individuals in the SSS and control conditions to complete outcome surveys and gather preliminary effectiveness data on the SSS intervention. Hypothesis 2a: Victims who disclose to an individual in the SSS intervention (n=50) will report trends towards receiving more positive social reactions to disclosure, less negative social reactions to disclosure, and fewer symptoms of PTSD, depression, drinking to cope, and negative alcohol-related consequences compared to individuals who disclose to an individual in the control condition (n=50).

ELIGIBILITY:
Inclusion Criteria:

* undergraduate student at University of New Hampshire
* read and understand English
* able to independently complete online surveys

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1268 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Hampshire, Durham, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention-Attend: This arm was invited to and attended the intervention, followed by a six-month follow-up evaluation.
  Supporting Survivors and Self: An Intervention for Social Supports of Survivors of Partner Abuse and Sexual Aggression (SSS): The SSS intervention consists of a two-hour session followed by a 90-minute booster session a month following the initial program session. The SSS intervention is delivered in groups of approximately 20 students facilitated by peer educators. The SSS intervention provides participants with specific information on the reasons why positive social reactions are important and negative social reactions can be harmful, examples of what to say and what not to say (including ways to promote healthy coping and discourage unhealthy coping, e.g., drinking to cope), opportunities for roleplay, and an emphasis on the importance of self-care and ways in which self-care can be balanced with the needs of IPV and SA victims.
- Wait-list Control: This arm was be invited to attend the intervention after a six-month follow-up evaluation.
- Intervention-Nonattend: This aim was invited to but did not attend the intervention, and completed the same six-month follow-up evaluation.
Period: Overall Study
Arm/Group | Intervention-Attend | Wait-list Control | Intervention-Nonattend
Started | 305 | 432 | 531
Completed | 261 | 314 | 314
Not Completed | 44 | 118 | 217
Not completed — Withdrawal by Subject | 44 | 118 | 217

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention-Attend | Wait-list Control | Intervention-Nonattend | Total
Number analyzed (Participants) | 305 | 432 | 531 | 1268
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 305 | 432 | 531 | 1268
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.50 (1.17) | 19.51 (1.27) | 19.64 (1.23) | 19.56 (1.23)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Woman | 239 | 276 | 351 | 866
  Man | 63 | 154 | 174 | 391
  Self-identify or No answer | 3 | 2 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 20 | 33 | 63
  Not Hispanic or Latino | 294 | 409 | 489 | 1192
  Unknown or Not Reported | 1 | 3 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 18 | 15 | 24 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 9 | 7 | 18
  White | 273 | 393 | 478 | 1144
  More than one race | 9 | 11 | 13 | 33
  Unknown or Not Reported | 2 | 3 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 305 | 432 | 531 | 1268

OUTCOME MEASURES:

1. Primary Outcome: Negative Social Reactions
Description: As measured by the Social Reactions Questionnaire (at six month follow-up). This scale is measured from 1 to 6, with higher mean scores representing a less desirable outcome.
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: Mean of actual negative reactions scale
Arm/Group | Intervention-Attend | Wait-list Control | Intervention-Nonattend
Number analyzed (Participants) | 130 | 164 | 159
Mean of actual negative reactions scale | 1.25 (0.37) | 1.28 (0.40) | 1.35 (0.56)

2. Secondary Outcome: Positive Social Reactions
Description: as for outcome 1
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention-Attend | Wait-list Control | Intervention-Nonattend
Number analyzed (Participants) | 129 | 160 | 158
score on a scale | 4.05 (0.68) | 3.87 (0.82) | 3.87 (0.74)

ADVERSE EVENTS:
Time Frame: Six months.
Description: No adverse events to report.
Arm/Group | Intervention-Attend | Wait-list Control | Intervention-Nonattend
All-Cause Mortality (participants affected / at risk) | 0/305 | 0/432 | 0/531
Serious Adverse Events (participants affected / at risk) | 0/305 | 0/432 | 0/531
Other Adverse Events (participants affected / at risk) | 0/305 | 0/432 | 0/531

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT03488927/Prot_001.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT03488927/SAP_002.pdf
  • Informed Consent Form (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT03488927/ICF_003.pdf